CLINICAL TRIAL: NCT01362686
Title: Comparative Effectiveness Research Trial of Alzheimer's Disease Drugs
Brief Title: Comparative Research of Alzheimer's Disease Drugs
Acronym: COMET-AD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low study accrual caused the study to be ended early.
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Malaz Boustani, MD, MPH, Regenstrief Institute, IU Center for Aging Reserach Scientist, Regenstrief Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HS019818-01 (AHRQ); R01HS019818-01 (AHRQ)
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: diagnosis of Alzheimer's disease; medication adherence
MeSH Terms: conditions — Dementia; Alzheimer Disease; Medication Adherence | interventions — Donepezil; Galantamine; Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Donepezil (Experimental): See intervention note.
  Interventions: Drug: Donepezil
- Galantamine (Experimental): See intervention note.
  Interventions: Drug: Galantamine
- Rivastigmine (Experimental): See intervention note.
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Donepezil — The study is open-label and the memory care practice physicians will make determinations about initial drug dosage and any dosage changes and the timing of those changes. These physicians will also make the determination about whether to switch to a different anti-dementia drug, add memantine, or any other agent. We will, of course, monitor the frequency and content of such changes in the natural course of patient care.
  Other Names: Aricept
  Arms: Donepezil
Drug: Galantamine — The study is open-label and the memory care practice physicians will make determinations about initial drug dosage and any dosage changes and the timing of those changes. These physicians will also make the determination about whether to switch to a different anti-dementia drug, add memantine, or any other agent. We will, of course, monitor the frequency and content of such changes in the natural course of patient care.
  Other Names: Razadyne
  Arms: Galantamine
Drug: Rivastigmine — The study is open-label and the memory care practice physicians will make determinations about initial drug dosage and any dosage changes and the timing of those changes. These physicians will also make the determination about whether to switch to a different anti-dementia drug, add memantine, or any other agent. We will, of course, monitor the frequency and content of such changes in the natural course of patient care.
  Other Names: Exelon
  Arms: Rivastigmine

SUMMARY:
Conduct a comparative effectiveness clinical trial of medication treatment for behavioral symptoms of Alzheimer's disease in a group of real-world memory care clinics with enhanced access to the Indiana Network for Patient Care.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to enhance the existing information technology infrastructure in Central Indiana to improve the nation's capacity to conduct comparative effectiveness research (CER). Consistent with the instructions in RFA-HS-10-005, the investigators propose to apply these new capacities to a novel CER project evaluating treatment for Alzheimer's disease. Alzheimer's disease has been identified as a first quartile CER priority. This proposal represents collaboration between the Medical Informatics Program at the Regenstrief Institute, Inc (a world leader in health information technology) and two Indiana University research programs: the Center for Aging Research and the Division of Clinical Pharmacology. These programs have an established track record in research relevant to under-served populations. Thus, this proposal combines considerable investigator, environment, and research strengths to continue to build a novel CER infrastructure in support of the nation's evidentiary CER priorities.

Throughout this proposal, the investigators use the AHRQ definition of CER: the conduct and synthesis of research comparing the benefits and harms of different interventions and strategies to prevent, diagnose, treat and monitor health conditions in real world settings." The investigators also refer to a clinical trial of medication treatment for behavioral symptoms of Alzheimer's disease as the specific CER proposed to demonstrate the potential of our new infrastructure. However, the investigators stress that the enhancements proposed to existing infrastructure would support a broad portfolio of CER across an array of priority conditions. The investigators are also proposing enhancements in our privacy and confidentiality technology that would allow researchers from across the country to access de-identified data in support of CER. In summary, the investigators are proposing to add new CER knowledge on Alzheimer' disease and thereby field test new information technology capacities important to a wide range of CER projects while also increasing our capacity to provide data and opportunities for nationwide CER.

The derivation of meaningful and actionable evidence from CER ultimately depends on capturing relevant, comprehensive and accurate data about treatment decisions, patients' clinical status, their care processes and environment, and the health outcomes they experience and value. Such data must be tracked longitudinally in order to determine temporal relationships, cause-effect paradigms, and the efficacy of specific clinical interventions in the context of other conditions, interventions, and goals of care. At Indiana University and the Regenstrief Institute, the investigators have four decades of experience and a well-documented, world-class clinical informatics and research infrastructure for capturing, storing, querying and analyzing treatment patterns and patients' clinical outcomes.

The maturation of this health information technology is now embodied within the Indiana Network for Patient Care (INPC), a fully-operational regional health information exchange. The investigators are well positioned to expand and leverage this infrastructure in support of local and national multi-site clinical trials in comparative effectiveness. The specific aims of this proposal are to:

1.0 PROSPECT STUDY: Enhance our existing information technology infrastructure to:

1. provide de-identified access to the INPC database for CER work
2. capture, store, and track a broader array of health care outcomes important to patients and their caregivers (e.g. behavioral symptoms due to dementia);
3. support providers' and caregivers' and researchers' increasing need to work in teams by providing new tools for communication and co-management (e.g. collaborative care and research)

2.0 COMET-AD STUDY: Conduct comparative effectiveness clinical trial of medication treatment for behavioral symptoms of Alzheimer's disease in a group of real-world memory care clinics with enhanced access to the Indiana Network for Patient Care.

ELIGIBILITY:
Inclusion Criteria:

* older adults with a diagnosis of possible or probable Alzheimer's disease
* planning to initiate treatment with a cholinesterase inhibitor
* planning to continue care in the memory care practice
* participation by a family caregiver willing to complete the study outcome assessments
* access to a telephone
* ability to understand English-Language survey instruments

Exclusion Criteria:

• prior serious adverse event from the study medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Regenstrief Institute, Center for Aging Research
Locations (5):
- United States (5):
  - Touchpoint, Fishers, Indiana
  - Methodist Center for Geriatric Medicine, Indianapolis, Indiana
  - University Clinical Neurology, Indianapolis, Indiana
  - Wishard Health Services, Indianapolis, Indiana
  - St. Vincent Center for Healthy Aging, Indianapolis, Indiana

REFERENCES:
- [Background] Callahan CM, Boustani MA, Unverzagt FW, Austrom MG, Damush TM, Perkins AJ, Fultz BA, Hui SL, Counsell SR, Hendrie HC. Effectiveness of collaborative care for older adults with Alzheimer disease in primary care: a randomized controlled trial. JAMA. 2006 May 10;295(18):2148-57. doi: 10.1001/jama.295.18.2148. PMID 16684985
- [Background] Boustani M, Callahan CM, Unverzagt FW, Austrom MG, Perkins AJ, Fultz BA, Hui SL, Hendrie HC. Implementing a screening and diagnosis program for dementia in primary care. J Gen Intern Med. 2005 Jul;20(7):572-7. doi: 10.1111/j.1525-1497.2005.0126.x. PMID 16050849
- [Background] Boustani MA, Frame A, Munger S, Healey P, Westlund J, Farlow M, Hake A, Austrom MG, Shepard P, Bubp C, Azar J, Nazir A, Adams N, Campbell NL, Chehresa A, Dexter P. Connecting research discovery with care delivery in dementia: the development of the Indianapolis Discovery Network for Dementia. Clin Interv Aging. 2012;7:509-16. doi: 10.2147/CIA.S36078. Epub 2012 Nov 16. PMID 23204843
- [Background] Campbell N, Boustani M, Limbil T, Ott C, Fox C, Maidment I, Schubert CC, Munger S, Fick D, Miller D, Gulati R. The cognitive impact of anticholinergics: a clinical review. Clin Interv Aging. 2009;4:225-33. doi: 10.2147/cia.s5358. Epub 2009 Jun 9. PMID 19554093
- [Derived] Lim AWY, Schneider L, Loy C. Galantamine for dementia due to Alzheimer's disease and mild cognitive impairment. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD001747. doi: 10.1002/14651858.CD001747.pub4. PMID 39498781
- [Derived] Campbell NL, Perkins AJ, Gao S, Skaar TC, Li L, Hendrie HC, Fowler N, Callahan CM, Boustani MA. Adherence and Tolerability of Alzheimer's Disease Medications: A Pragmatic Randomized Trial. J Am Geriatr Soc. 2017 Jul;65(7):1497-1504. doi: 10.1111/jgs.14827. Epub 2017 Mar 14. PMID 28295141
- [Derived] Campbell NL, Dexter P, Perkins AJ, Gao S, Li L, Skaar TC, Frame A, Hendrie HC, Callahan CM, Boustani MA. Medication adherence and tolerability of Alzheimer's disease medications: study protocol for a randomized controlled trial. Trials. 2013 May 4;14:125. doi: 10.1186/1745-6215-14-125. PMID 23782591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from 2011-2014. Recruitment took place in geriatric and memory care specialty clinics in an urban setting. Registered nurses, nurse practitioners, and research assistants completed the recruitment and informed consent procedures.
Pre-assignment Details: The enrollment goal in the original protocol of the study was 200 patient-caregiver dyads. 200 were enrolled, but it was discovered that 4 dyads were ineligible after enrollment and were not randomized or included in the study which brings the total enrollment to 196. Recruitment was then terminated due to low enrollment rate.
Period: Overall Study
Arm/Group | Donepezil | Galantamine | Rivastigmine
Started | 67 | 66 | 63
Completed | 59 | 54 | 53
Not Completed | 8 | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Galantamine | Rivastigmine | Total
Number analyzed (Participants) | 67 | 66 | 63 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.1 (7.6) | 80.1 (9.6) | 81.6 (7.8) | 80.2 (8.4)
Gender [Count of Participants; unit: Participants]
  Female | 19 | 20 | 12 | 51
  Male | 48 | 46 | 51 | 145

OUTCOME MEASURES:

1. Primary Outcome: Discontinuation Rates
Description: We are not seeking to establish efficacy of these three medications for the indication of Alzheimer's disease. Each of these medications already has FDA-approval for Alzheimer's. The primary outcome measure is the discontinuation rate among the three medications. Based on previous systematic reviews, these rates are reportedly in the range of 30% by 12 weeks compared with placebo. We will determine the approximate date of discontinuation by self-reports from the caregiver through the telephone-based interview at 6, 12, and 18 weeks.
Time Frame: 6, 12, and 18 week interviews from enrollment
Measure: Number; unit: participants
Arm/Group | Donepezil | Galantamine | Rivastigmine
Number analyzed (Participants) | 67 | 66 | 63
participants | 26 | 35 | 37

2. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: The NPI is based on a structured interview administered to an informal caregiver and has been adopted by the Alzheimer's Disease Cooperative Studies Group to obtain information on the presence of psychopathology in behavioral areas including delusions, apathy, hallucinations, disinhibition, agitation, depression, aberrant motor behavior, anxiety, night-time behavior, and euphoria.9 For each of 12 symptoms, if the caregiver reports the presence of psychopathology, a frequency and severity score are multiplied to yield a possible item score range of 0-12, and a possible total score range of 0-144. The NPI can be used to assess changes in the patient's behavior over the past month. The NPI also assesses the level of caregiver distress attributable to each of the 12 patient behaviors, with a possible total caregiver distress score range of 0-60. Higher scores indicate higher severity of psychopathology and caregiver disress. The NPI has excellent reliability and validity.
Time Frame: Baseline, 6, 12, 18 week interviews from enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil | Galantamine | Rivastigmine
Number analyzed (Participants) | 59 | 58 | 54
units on a scale
  6 WeekNPI Patient | 12.71 (17.10) | 9.42 (13.21) | 8.63 (11.73)
  6 Week NPI Caregiver | 5.94 (9.09) | 4.40 (5.80) | 3.91 (4.86)
  12 Week NPI Patient | 9.62 (13.56) | 8.40 (13.27) | 5.24 (5.54)
  12 Week NPI Caregiver | 5.66 (7.34) | 4.33 (6.01) | 2.22 (2.86)
  18 Week NPI Patient | 9.06 (13.87) | 10.67 (13.85) | 7.26 (7.36)
  18 Week NPI Caregiver | 5.56 (7.66) | 6.22 (7.56) | 2.89 (3.17)

3. Secondary Outcome: Healthy Aging Brain Care (HABC)-Monitor
Description: The current HABC-Monitor includes 30 items covering four clinically relevant domains of dementia, ie, cognitive, functional, behavioral, and psychological symptoms, and caregiver quality of life. For brevity and practical use in the clinical setting, each item on the four scales was designed to have the same item response options consisting of four categories that use the frequency of the target problem in the past 2 weeks. The HABC- Monitor took approximately 6 minutes to complete. The scores of the four scales are summed to create the total scores which were used in this analysis.The higher the total score, the higher the level of self reported caregiver burden. The minimum score is 0 and the maximum score is 90.
Time Frame: baseline, 6, 12, and 18 week interviews
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil | Galantamine | Rivastigmine
Number analyzed (Participants) | 59 | 58 | 54
units on a scale
  Baseline HABC | 18.76 (13.64) | 18.34 (11.91) | 16.61 (11.49)
  6 Week HABC | 18.61 (15.16) | 19.16 (12.72) | 16.43 (10.52)
  12 Week HABC | 16.04 (13.41) | 18.00 (15.71) | 13.63 (9.34)
  18 Week HABC | 16.90 (15.30) | 19.92 (14.28) | 15.80 (9.01)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 6 weeks, 12 weeks, and 18 weeks.
Arm/Group | Donepezil | Galantamine | Rivastigmine
Serious Adverse Events (participants affected / at risk) | 32/59 | 29/54 | 27/53
Other Adverse Events (participants affected / at risk) | 40/59 | 42/54 | 35/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=59) | Galantamine (N=54) | Rivastigmine (N=53)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 2 (2)
Diahrrhea (Gastrointestinal disorders) | 13 (17) | 5 (5) | 7 (8)
Dizziness (Nervous system disorders) | 4 (4) | 6 (10) | 8 (9)
Fainting (General disorders) | 2 (2) | 1 (1) | 2 (2)
Falls (General disorders) | 0 (0) | 0 (0) | 3 (3)
Fast or Slowed Heart Rate (Cardiac disorders) | 5 (7) | 0 (0) | 4 (5)
Feeling Tired (General disorders) | 7 (10) | 5 (7) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 4 (6) | 3 (4)
Incontinence (General disorders) | 5 (6) | 6 (9) | 5 (6)
Irregular Heart Beat (Cardiac disorders) | 4 (4) | 3 (4) | 3 (3)
Lack of Interest in Eating (Metabolism and nutrition disorders) | 9 (10) | 3 (3) | 4 (4)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (8) | 3 (5)
Nightmares (Psychiatric disorders) | 6 (8) | 3 (5) | 1 (1)
Pain (Nervous system disorders) | 3 (5) | 7 (10) | 4 (5)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (6) | 4 (4)
Seizure or Fits (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=59) | Galantamine (N=54) | Rivastigmine (N=53)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 2 (2)
Diahrrhea (Gastrointestinal disorders) | 11 (12) | 13 (16) | 9 (9)
Dizziness (General disorders) | 13 (14) | 12 (16) | 9 (9)
Fainting (General disorders) | 5 (6) | 2 (2) | 1 (1)
Falls (General disorders) | 6 (7) | 5 (6) | 4 (4)
Fast or Slowed Heart Rate (Cardiac disorders) | 5 (6) | 4 (5) | 0 (0)
Feeling Tired (General disorders) | 15 (21) | 17 (24) | 14 (16)
Headache (Nervous system disorders) | 4 (4) | 9 (10) | 4 (6)
Incontinence (General disorders) | 10 (14) | 10 (12) | 9 (13)
Irregular Heart Beat (Cardiac disorders) | 3 (4) | 5 (5) | 1 (1)
Lack of Interest in Eating (Metabolism and nutrition disorders) | 12 (12) | 7 (8) | 12 (15)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (6) | 5 (10)
Nightmares (Psychiatric disorders) | 7 (8) | 5 (7) | 1 (1)
Pain (Nervous system disorders) | 6 (6) | 6 (6) | 6 (6)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 13 (18) | 8 (9)
Seizure or Fits (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size limits generalizability and may introduce type II error. The study took place at a time when most third-party payers declared donepezil the preferred AChEI due to cost that may have influenced study's results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No